CLINICAL TRIAL: NCT04861168
Title: Driving Pressure Guided Ventilation Versus Conventional Lung Protective Strategy in Morbid Obese Patients Undergoing Laparoscopic Bariatric Surgery; a Prospective Randomized Controlled Study
Brief Title: Driving Pressure Guided Ventilation Versus Conventional Lung Protective Strategy in Morbid Obese Patients Undergoing Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Saed Aly Elbehairy, Assisstant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Driving pressure ventilation
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Driving Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Driving pressure guided ventilation (Experimental): Patients will be mechanically ventilated with driving pressure guided ventilation with VT 6-8 ml /kg of predicted body weight, and after recruitment we will return to the baseline PEEP 5 cmH2O that will be increased by 2 cmH2O until reaching the lowest possible driving pressure for every patient. Each PEEP level will be applied for 10 respiratory cycles and DP will be calculated at the last cycle.
  Interventions: Procedure: driving pressure guided ventilation
- Conventional protective lung strategy (Active Comparator): Patients will be mechanically ventilated with conventional protective lung strategy with VT 6-8 ml /kg of predicted body weight, after recruitment, we will return to the baseline PEEP 5 cmH2O and will be maintained until the end of surgery.
  Interventions: Procedure: Conventional protective lung strategy

INTERVENTIONS:
Procedure: driving pressure guided ventilation — driving pressure guided ventilation
  Arms: Driving pressure guided ventilation
Procedure: Conventional protective lung strategy — Conventional protective lung strategy
  Arms: Conventional protective lung strategy

SUMMARY:
This study will be conducted to evaluate the effect of driving pressure guided ventilation compared with conventional protective lung ventilation during laparoscopic bariatric surgeries in morbid obese patients.

* the primary outcome: Intraoperative oxygenation measured by the arterial partial pressure of oxygen (PaO2).
* the secondary outcome: incidence of early postoperative pulmonary complications e.g., postoperative hypoxia, the need for supplementary oxygen, atelectasis, barotrauma, and respiratory failure.

DETAILED DESCRIPTION:
Protective mechanical ventilation during anesthesia aims at minimizing lung injury and has been associated to a decrease in postoperative pulmonary complications (PPCs). Conventional protective ventilation strategy is consisted of the use of a low tidal volume (VT) and fixed moderate positive end expiratory pressure (peep). However, low-VT may result in the reduction of the functional volume of the lung manifested as lung collapse. Another potential consequence of lung collapse is the impairment in ventilatory efficiency.

Bariatric surgery is proven to achieve significant and sustained weight loss in the morbidly obese. Major weight loss can lead to partial/complete resolution of a range of conditions including, diabetes mellitus, ischemic heart disease, and hypertension.

Obese patients undergoing general anesthesia and mechanical ventilation during abdominal and bariatric surgeries commonly have a higher incidence of postoperative pulmonary complications (PPCs), due to factors such as decreasing oxygen reserve, declining functional residual capacity, and reducing lung compliance. And also pneumoperitoneum aggravates pulmonary atelectasis caused by mechanical ventilation, especially in obese patients.

Driving pressure (DP) which is the difference between the airway pressure at the end of inspiration (plateau pressure, (Ppl) and PEEP was first introduced by Amato et al in 2015 in their meta-analy¬sis study for ARDS patients. The authors suggested that driving pressure is the stronger predictor of mortality as compared with low VT and Ppl.

Several retrospec¬tive and prospective studies confirmed the importance of driving pressure in ARDS pa¬tients and during general anesthesia without differentiation between obese and nonobese patients .only one retrospective study showed that driving pressure was not associated with mortality in obese-ARDS patients. we hypothesize that these results may be different in obese patients having healthy lungs.

ELIGIBILITY:
Inclusion Criteria:

* sixty patients have a BMI 40-50 kg/m2, ASA physical status III, aged between 18 and 60 years, scheduled to undergo laparoscopic bariatric surgeries.

Exclusion Criteria:

* patient refusal to participate in the study.
* Patients had a recent history of severe respiratory disease and previous major pulmonary surgeries.
* patients who are contraindicated with application of PEEP (high intracranial pressure, bronchopleural fistula, hypovolemic shock, right ventricular failure).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative oxygenation measured by the arterial partial pressure of oxygen (PaO2). | the time of surgery
  Arterial blood gases -for measurement of pao2- will be sampled after induction of anesthesia (baseline) ,10 minutes after recruitment, before end of surgery, and 30 minutes after extubation.

SECONDARY OUTCOMES:
the need for rescue recruitment | the time of surgery
  the need for rescue recruitment
incidence of early postoperative pulmonary complications e.g., postoperative hypoxia, the need for supplementary oxygen, atelectasis, barotrauma, and respiratory failure. | First 24 hours postoperative
  ncidence of early postoperative pulmonary complications e.g., postoperative hypoxia, the need for supplementary oxygen, atelectasis, barotrauma, and respiratory failure.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Tanta University Hospitals, Tanta
  - Faculty of Medicine, Tanta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Biehl M, Binnekade JM, Canet J, Fernandez-Bustamante A, Futier E, Gajic O, Hedenstierna G, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Putensen C, Ranieri M, Scavonetto F, Schilling T, Schmid W, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network Investigators. Protective versus Conventional Ventilation for Surgery: A Systematic Review and Individual Patient Data Meta-analysis. Anesthesiology. 2015 Jul;123(1):66-78. doi: 10.1097/ALN.0000000000000706. PMID 25978326
- [Background] Unzueta C, Tusman G, Suarez-Sipmann F, Bohm S, Moral V. Alveolar recruitment improves ventilation during thoracic surgery: a randomized controlled trial. Br J Anaesth. 2012 Mar;108(3):517-24. doi: 10.1093/bja/aer415. Epub 2011 Dec 26. PMID 22201185
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Derived] Elbehairy MS, Eid GM, Elzeftawy AE, Elsheikh NA, Messbah WE. Driving pressure guided ventilation versus conventional lung protective strategy in morbid obese patients undergoing laparoscopic bariatric surgery: a prospective randomized controlled study. BMC Anesthesiol. 2025 Nov 20;25(1):577. doi: 10.1186/s12871-025-03431-1. PMID 41266983